CLINICAL TRIAL: NCT00719264
Title: A Randomized, Open-label, Multi-center Phase II Study to Compare Bevacizumab Plus RAD001 Versus Interferon Alfa-2a Plus Bevacizumab for the First-line Treatment of Patients With Metastatic Clear Cell Carcinoma of the Kidney
Brief Title: Safety and Efficacy of Bevacizumab Plus RAD001 Versus Interferon Alfa-2a and Bevacizumab for the First-line Treatment in Adult Patients With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001L2201; 2008-000077-38 (EudraCT Number)
Record Dates: First submitted 2008-07-15; First posted 2008-07-21 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma; Adenocarcinoma; Renal Cell; Nephroid Carcinoma; Hypernephroid
Keywords: Renal cell carcinoma; Adults; Bevacizumab; RAD001; Everolimus; Interferon; Clear; Roferon; Avastin; Nephrectomy; newly diagnosed
MeSH Terms: conditions — Carcinoma; Adenocarcinoma; Carcinoma, Renal Cell; Margins of Excision | interventions — Everolimus; Interferon alpha-2; Bevacizumab

ARMS (2):
- bevacizumab, RAD001 (everolimus) (Experimental): Participants received oral everolimus 10 mg qd plus intravenous bevacizumab 10mg/kg every 2 weeks
  Interventions: Drug: RAD001(everolimus); Drug: bevacizumab
- bevacizumab, interferon alfa-2a (IFN) (Active Comparator): Participants received subcutaneous IFN dose escalated from 3 MIU (million international unit) during week 1, 6 MIU during week 2, and 9 MIU during week 3 of treatment and subsequently (if tolerated), 3 times per week plus intravenous bevacizumab 10 mg/kg every 2 weeks
  Interventions: Drug: interferon alfa-2a; Drug: bevacizumab

INTERVENTIONS:
Drug: RAD001(everolimus) — 10 mg qd
  Other Names: Afinitor
  Arms: bevacizumab, RAD001 (everolimus)
Drug: interferon alfa-2a — dose escalated from 3 MIU (million international unit) during week 1, 6 MIU during week 2, and 9 MIU during week 3
  Arms: bevacizumab, interferon alfa-2a (IFN)
Drug: bevacizumab — 10 mg/kg every 2 weeks

SUMMARY:
To estimate the difference in efficacy and safety of bevacizumab and RAD001 compared to bevacizumab and interferon alfa-2a for first-line treatment of patients with metastatic carcinoma of the kidney.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic renal cell carcinoma
2. Patients with at least one measurable lesion
3. Patients with progressive metastatic renal cell carcinoma
4. Patients who had a prior partial or complete nephrectomy
5. Patients with a Karnofsky Performance Status ≥70%.
6. Adequate bone marrow function
7. Adequate liver function
8. Adequate renal function
9. Adequate coagulation profile

Exclusion Criteria:

1. 4 weeks post-major surgery
2. Patients who had radiation therapy within 28 days prior to start of study
3. Patients in need for major surgical procedure during the course of the study.
4. Patients with a serious non-healing wound, ulcer, or bone fracture.
5. Patients with a history of seizure(s) not controlled with standard medical therapy.
6. Patients who have received prior systemic treatment for their metastatic RCC.
7. Patients who received prior therapy with VEGF pathway inhibitor
8. Patients who have previously received systemic mTOR inhibitors
9. Patients with a known hypersensitivity RAD001 (everolimus) or other rapamycins or to its excipients.
10. Patients with history or current central nervous system (CNS) metastases or spinal cord compression.
11. Patients with a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
12. Patients with proteinuria at screening.
13. Patients with inadequately controlled hypertension
14. Patients receiving ongoing or with recent need for full therapeutic dose of oral or parenteral anticoagulants or chronic daily treatment with aspirin
15. Patients receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent.
16. Patients with a known history of HIV
17. Patients with hypersensitivity to interferon alfa-2a or any component of the product.
18. Patients with an active, bleeding diathesis or coagulopathy or recurrent thromboembolism
19. Patients who have any severe and/or uncontrolled medical conditions or other conditions
20. Left Ventricular Ejection Fraction < lower limit of institutional normal assessed by ECHO or MUGA
21. Patients who have a history of another primary malignancy ≤ 3 years
22. Female patients who are pregnant or breast feeding
23. Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study treatment start.
24. Patients unwilling to or unable to comply with the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2008-11-12 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2013-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (99):
- United States (9):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - City of Hope National Medical Center Dept.ofCityofHopeMedicalCtr(3), Duarte, California
  - USC/Kenneth Norris Comprehensive Cancer Center Regulatory Contact 3, Los Angeles, California
  - University of California at Los Angeles Dept. of Hem/Oncology, Los Angeles, California
  - Karmanos Cancer Institute Dept.of KarmanosCancerInst (5), Detroit, Michigan
  - Nevada Cancer Institute Dept. of Nevada Cancer (3), Las Vegas, Nevada
  - St. Luke's Hospital and Health Network St. Luke's Cancer Network, Bethlehem, Pennsylvania
  - Las Colinas Hematology Oncology Grapevine, Irving, Texas
  - Seattle Cancer Care Alliance Dept. of SCCA, Seattle, Washington
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (5):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Egypt (2):
  - Novartis Investigative Site, Cairo, Egypt
  - Novartis Investigative Site, Cairo
- France (12):
  - Novartis Investigative Site, Strasbourg, Cedex
  - Novartis Investigative Site, Suresnes, France
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Montellier Cedex 5
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Tübingen
- Hong Kong (2):
  - Novartis Investigative Site, Shatin, New Territories, Hong Kong
  - Novartis Investigative Site, Tuenmen, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Italy (13):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Trento, TN
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Leiden, Netherlands, Netherlands
- Russia (4):
  - Novartis Investigative Site, Moscow, Moscow
  - Novartis Investigative Site, Obninsk, Russia
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- South Africa (2):
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Pretoria
- South Korea (5):
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (6):
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Zaragoza, Zaragoza
  - Novartis Investigative Site, Santander
- Switzerland (2):
  - Novartis Investigative Site, Bern, Switzerland
  - Novartis Investigative Site, Chur
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Linkou District
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Adana, Turkey
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Bursa, Turkey
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Mecidiyekoy/Istanbul
- United Kingdom (3):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Ravaud A, Barrios CH, Alekseev B, Tay MH, Agarwala SS, Yalcin S, Lin CC, Roman L, Shkolnik M, Anak O, Gogov S, Pelov D, Louveau AL, Melichar B. RECORD-2: phase II randomized study of everolimus and bevacizumab versus interferon alpha-2a and bevacizumab as first-line therapy in patients with metastatic renal cell carcinoma. Ann Oncol. 2015 Jul;26(7):1378-84. doi: 10.1093/annonc/mdv170. Epub 2015 Apr 7. PMID 25851632
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/etrials/searchTrial.do?t=i&trialID=688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Started | 182 | 183
Full Analysis Set | 182 | 183
Safety Set | 180 | 181
Completed | 0 | 0
Not Completed | 182 | 183
Not completed — Adverse Event | 41 | 49
Not completed — Death | 13 | 10
Not completed — Administrative Problems | 6 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Protocol Deviation | 1 | 3
Not completed — New Cancer Therapy | 4 | 2
Not completed — Disease Progression | 104 | 107

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN) | Total
Number analyzed (Participants) | 182 | 183 | 365
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.71 (10.584) | 59.93 (10.272) | 60.32 (10.422)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 52 | 96
  Male | 138 | 131 | 269

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) of Participants Who Received RAD001 Plus Bevacizumab Versus Participants Who Received IFN Plus Bevacizumab
Description: Tumor response and disease progression were assessed using response evaluation criteria in solid tumors (RECIST), version 1.0. All target and non-target lesions identified at baseline were assessed using the same method, CT scan with contrast or MRI with contrast, throughout the trial. All scans were reviewed by independent, central radiology. Disease progression was defined as: 1) a 20% increase in the sum of the longest diameter of all target lesions, taking as reference the smallest sum of the longest diameters of all target lesions recorded at or after baseline or 2) the appearance of a new lesions or 3) the unequivocal progression of non-target lesions overall.
Time Frame: Time from randomization to the date of radiological progressive disease as per independent central review, death from any cause, or last tumor assessment, reported between date of first participant randomized until 31Dec2011, cutoff date.
Population: Full Analysis Set: This set consists of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 182 | 183
Months | 9.3 [8.1 to 11.2] | 10.0 [8.3 to 12.9]

2. Secondary Outcome: Overall Survival (OS) Treatment Effect in Participants Who Received RAD001 Plus Bevacizumab Versus Participants Who Received IFN Plus Bevacizumab
Description: Overall survival (OS) was defined as the time of randomization to the date of death due to any cause.
Time Frame: Time from randomization to the date of death from any cause, reported between date of first participant randomized and up to 2 years after the last participant randomized (data cutoff: 30Aug2012)
Population: Full Analysis Set: This set consists of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 182 | 183
Months | 27.1 [19.9 to 35.3] | 27.1 [20.4 to 30.8]

3. Secondary Outcome: Best Overall Response in Participants Who Received RAD001 Plus Bevacizumab Versus Participants Who Received IFN Plus Bevacizumab
Description: Overall response is defined as the number of participants having achieved confirmed Complete Response (CR) + Partial Response (PR). Confirmed CR = at least two determinations of CR at least 4 weeks apart before progression. Confirmed PR = at least two determinations of PR or better at least 4 weeks apart before progression. CR required a disappearance of all target and non-target lesions. PR required at least a 30% decrease in the sum of the longest diameters of all target lesions, taking as a reference the baseline sum of the longest diameters. Disease progression was defined as: 1) a 20% increase in the sum of the longest diameter of all target lesions, taking as reference the smallest sum of the longest diameters of all target lesions recorded at or after baseline or 2) the appearance of a new lesions or 3) the unequivocal progression of non-target lesions overall.
Time Frame: Time from first participant randomized until 31Dec2011, cutoff date.
Population: Full Analysis Set: This set consists of all randomized participants.
Measure: Number; unit: Number of participants
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 182 | 183
Number of participants
  Complete response (CR) | 0 | 1
  Partial response (PR) | 49 | 50
  Stable disease (SD) | 90 | 84
  Progressive disease (PD) | 25 | 26
  Unknown response | 18 | 22
  Overall objective response (CR+PR) | 49 | 51

4. Secondary Outcome: Response Duration Differences in Participants Who Received RAD001 Plus Bevacizumab Versus Participants Who Received IFN Plus Bevacizumab
Description: The duration of response, applied only to participants with best overall response at CR or PR, is defined as the number of days between the date of first documented response (CR or PR) and the date of the event: radiological progression as per central review or death due to underlying cancer, whichever occurs first. If no event, participant is censored at the last adequate assessment.
Time Frame: Time from first documented response date of radiological progressive disease as per independent central review, death due to underlying cancer, or last tumor assessment, reported between date of first participant randomized until 31Dec2011, cut-off date.
Population: A subset of participants from the full analysis set were analyzed. The full analysis set consists of all randomized participants. the subset includes participants who were complete responders or partial responders.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 49 | 51
Months | 13.3 [10.7 to 16.7] | 11.3 [10.4 to NA] — The upper limit was not estimable as it is longer than the estimated time period per data cutoff (31Dec2011).

5. Secondary Outcome: Number of Participants Who Experienced Adverse Events (AEs), Serious Adverse Events and Deaths
Description: Participants were monitored for adverse events, serious adverse events and deaths throughout the study. Participants were assessed continuously at each 28-day cycle.
Time Frame: From the first participant randomized until the last patient discontinued the study treatment + 28 days
Population: Safety Set: The safety set included all participants who received at least one dose of study drug (everolimus, bevacizumab or IFN) and had a valid post-baseline assessment. No AE or occurrence of death, noted at assessment, constitutes a valid post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 180 | 181
Participants
  Adverse events (serious and non-serious) | 179 | 180
  Serious adverse events | 79 | 76
  Deaths | 93 | 95

6. Secondary Outcome: Time to Definitive Deterioration of the Functional Assessment of Cancer Therapy Kidney Symptom Index, Disease Related Symptoms (FKSI-DRS) Risk Score by at Least 2 Score Units
Description: The analysis of this outcome measure was based on the FKSI-DRS scale which is a validated disease-related symptom index containing 9 items that measure symptoms predominantly related to kidney cancer. Each item is scored on a 5-point scale (0 = not at all; 4 = very much). If at least 5 of the 9 questions have been answered, the FKSI-DRS total score is calculated by subtracting nine times the mean of the scores of the answered items from 36. Participants with less than 5 out of the 9 questions answered will have a missing FKSI-DRS total score. The FKSI-DRS total score ranges from 0 (most severe symptoms) to 36 (no symptoms). Definitive deterioration is defined as a decrease by at least 2 units compared to baseline, with no later increase above this threshold observed during the study. A single measure reporting a decrease of at least 2 units was considered definitive only if it is the last one available for the participant.
Time Frame: Time from randomization to the date of definitive deterioration (defined as no later increase above the threshold observed during the study), or date of last assessment, reported between date of first patient randomized until 31Dec2011
Population: Full Analysis Set: This set consists of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 182 | 183
Months | 7.4 [4.7 to 10.8] | 8.0 [3.7 to 11.5]

7. Secondary Outcome: Time to Definitive Deterioration of the Global Health Status and the Physical Functioning (PF) Subscale Scores of the European Organization for the Research and Treatment of Cancer (EORTC)-Core Quality of Life Questionnaire (QLQ-C30) by at Least 10%
Description: The EORTC QLQ-C30 contains 30 items. These include five functional scales (physical, role, emotional, social and cognitive functioning), three symptom scales (fatigue, pain, nausea, and vomiting), a global health status/QoL scale, and six single items (dyspnea, diarrhea, constipation, anorexia, insomnia and financial impact). The PF subscale consists of 5 questions each scored from 1 (not at all) to 4 (very much). The score for the PF subscale and global health status range from 0 to 100, with a higher score representing a high level of functioning/high quality of life. Definitive deterioration by at least 10% is defined as a decrease in score by at least 10% compared to baseline, with no later increase above this threshold observed during the course of the study. A single measure reporting a decrease of at least 10% is considered definitive only if it is the last one available for the participant.
Time Frame: Time from randomization to the date of definitive deterioration (defined as no later increase above the threshold observed during the study), or date of last assessment, reported between date of first participant randomized until 31Dec2011
Population: Full Analysis Set: This set consists of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Number analyzed (Participants) | 182 | 183
Months
  Global health status/QoL | 7.4 [5.3 to 12.0] | 7.8 [5.6 to 10.2]
  Physical functioning | 8.5 [5.6 to 13.8] | 9.0 [6.5 to 12.9]

8. Secondary Outcome: Duration of Exposure of RAD001 in Participants Randomized to the Treatment Combination of RAD001 and Bevacizumab
Description: This outcome measure was assessed continuously.
Time Frame: From the date of the first participant treated until the last patient discontinued the study treatment + 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: weeks
Arm/Group | Bevacizumab, RAD001 (Everolimus)
Number analyzed (Participants) | 180
weeks | 37.0 [2 to 190]

ADVERSE EVENTS:
Arm/Group | Bevacizumab, RAD001 (Everolimus) | Bevacizumab, Interferon Alfa-2a (IFN)
Serious Adverse Events (participants affected / at risk) | 79/180 | 76/181
Other Adverse Events (participants affected / at risk) | 173/180 | 179/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, RAD001 (Everolimus) (N=180) | Bevacizumab, Interferon Alfa-2a (IFN) (N=181)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 2
CARDIAC FAILURE (Cardiac disorders) | 3 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 2 | 0
COLITIS (Gastrointestinal disorders) | 0 | 2
DIARRHOEA (Gastrointestinal disorders) | 5 | 1
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
ENTERITIS (Gastrointestinal disorders) | 1 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 1
GASTRIC FISTULA (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 4 | 2
PANCREATITIS (Gastrointestinal disorders) | 1 | 1
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 1 | 0
PROCTITIS (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
RETROPERITONEUM CYST (Gastrointestinal disorders) | 1 | 0
SIGMOIDITIS (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 3 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 4 | 2
ASTHENIA (General disorders) | 1 | 2
DISEASE PROGRESSION (General disorders) | 1 | 3
DRUG INEFFECTIVE (General disorders) | 0 | 1
FATIGUE (General disorders) | 2 | 3
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 | 4
GENERALISED OEDEMA (General disorders) | 1 | 0
HYPERPYREXIA (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 0
PYREXIA (General disorders) | 3 | 0
SUDDEN DEATH (General disorders) | 1 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
HEPATOTOXICITY (Hepatobiliary disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 3 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
INJECTION SITE INFECTION (Infections and infestations) | 0 | 1
LARYNGITIS (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 1
MYELITIS (Infections and infestations) | 0 | 1
NECROTISING FASCIITIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 1
PHARYNGITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 6 | 2
PYELONEPHRITIS (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
SEPSIS (Infections and infestations) | 4 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SINUSITIS BACTERIAL (Infections and infestations) | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 0
TUBERCULOSIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 3
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
CEMENT EMBOLISM (Injury, poisoning and procedural complications) | 1 | 0
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATINE INCREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 3 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 2
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 3
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 3
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 5
BONE LOSS (Musculoskeletal and connective tissue disorders) | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 3
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 3
COMA (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 1 | 1
DIZZINESS (Nervous system disorders) | 1 | 1
ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 2
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 2
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 2
DELIRIUM (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
SOPOR (Psychiatric disorders) | 0 | 1
BLADDER DILATATION (Renal and urinary disorders) | 0 | 1
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 1
OLIGURIA (Renal and urinary disorders) | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 1 | 2
RENAL COLIC (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 5 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 2
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACCELERATED HYPERTENSION (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 4 | 3
HYPERTENSIVE CRISIS (Vascular disorders) | 2 | 2
HYPOTENSION (Vascular disorders) | 1 | 0
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, RAD001 (Everolimus) (N=180) | Bevacizumab, Interferon Alfa-2a (IFN) (N=181)
ANAEMIA (Blood and lymphatic system disorders) | 35 | 35
LEUKOPENIA (Blood and lymphatic system disorders) | 4 | 12
LYMPHOPENIA (Blood and lymphatic system disorders) | 4 | 11
NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 21
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 | 29
TACHYCARDIA (Cardiac disorders) | 9 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 18 | 19
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 | 9
CONSTIPATION (Gastrointestinal disorders) | 30 | 26
DIARRHOEA (Gastrointestinal disorders) | 71 | 47
DRY MOUTH (Gastrointestinal disorders) | 3 | 11
DYSPEPSIA (Gastrointestinal disorders) | 8 | 11
GINGIVAL BLEEDING (Gastrointestinal disorders) | 3 | 11
MOUTH ULCERATION (Gastrointestinal disorders) | 13 | 3
NAUSEA (Gastrointestinal disorders) | 38 | 50
STOMATITIS (Gastrointestinal disorders) | 111 | 42
TOOTHACHE (Gastrointestinal disorders) | 16 | 12
VOMITING (Gastrointestinal disorders) | 25 | 26
ASTHENIA (General disorders) | 39 | 62
CHILLS (General disorders) | 4 | 21
FATIGUE (General disorders) | 57 | 75
INFLUENZA LIKE ILLNESS (General disorders) | 5 | 32
MALAISE (General disorders) | 2 | 11
OEDEMA PERIPHERAL (General disorders) | 44 | 18
PYREXIA (General disorders) | 24 | 63
GINGIVITIS (Infections and infestations) | 10 | 7
INFLUENZA (Infections and infestations) | 10 | 5
SINUSITIS (Infections and infestations) | 10 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 7
URINARY TRACT INFECTION (Infections and infestations) | 16 | 16
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 | 4
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 | 5
BLOOD CREATININE INCREASED (Investigations) | 20 | 7
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 10 | 13
WEIGHT DECREASED (Investigations) | 51 | 58
DECREASED APPETITE (Metabolism and nutrition disorders) | 48 | 80
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 40 | 8
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 18 | 5
HYPERKALAEMIA (Metabolism and nutrition disorders) | 5 | 11
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 24 | 17
HYPERURICAEMIA (Metabolism and nutrition disorders) | 3 | 14
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33 | 37
BACK PAIN (Musculoskeletal and connective tissue disorders) | 22 | 26
BONE PAIN (Musculoskeletal and connective tissue disorders) | 8 | 10
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 9 | 11
MYALGIA (Musculoskeletal and connective tissue disorders) | 11 | 34
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 25 | 17
DIZZINESS (Nervous system disorders) | 11 | 12
DYSGEUSIA (Nervous system disorders) | 21 | 7
HEADACHE (Nervous system disorders) | 36 | 38
DEPRESSION (Psychiatric disorders) | 8 | 25
INSOMNIA (Psychiatric disorders) | 23 | 25
DYSURIA (Renal and urinary disorders) | 10 | 10
PROTEINURIA (Renal and urinary disorders) | 90 | 68
COUGH (Respiratory, thoracic and mediastinal disorders) | 54 | 34
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 11 | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 28 | 32
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 62 | 38
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 18 | 7
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 12 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 13 | 9
DERMATITIS (Skin and subcutaneous tissue disorders) | 13 | 2
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 9 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 22 | 16
PRURITUS (Skin and subcutaneous tissue disorders) | 31 | 22
RASH (Skin and subcutaneous tissue disorders) | 42 | 20
HYPERTENSION (Vascular disorders) | 67 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.